CLINICAL TRIAL: NCT02244866
Title: A Randomized Controlled Trial to Compare the Efficacy Between Pergoveris and Follitropin Alfa in Ovarian Stimulation in Patients Aged ≥ 35 Years
Brief Title: Efficacy of Pergoveris in Aged IVF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_01_2012
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: IVF; LH supplementation; ovarian stimulation; poor responder
MeSH Terms: conditions — Infertility | interventions — pergoveris; Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pergoveris (FSH and LH) (Active Comparator): 150 IU of recombinant FSH and 75 IU of recombinant LH (Pergoveris) daily subcutaneous injection
  Interventions: Drug: Pergoveris (FSH and LH)
- Follitropin alpha (FSH) (Active Comparator): 150 IU of recombinant FSH (follitropin alpha or Gonal-F) daily subcutaneous injection
  Interventions: Drug: Follitropin alpha (FSH)

INTERVENTIONS:
Drug: Pergoveris (FSH and LH) — Drugs are injected subcutaneously everyday until ovarian follicles reach 17mm in diameter.
  Other Names: Pergoveris
  Arms: Pergoveris (FSH and LH)
Drug: Follitropin alpha (FSH) — Drugs are injected subcutaneously everyday until ovarian follicles reach 17mm in diameter.
  Other Names: Gonal-F
  Arms: Follitropin alpha (FSH)

SUMMARY:
To compare the efficacy between LH supplementation (Pergoveris) and non-LH supplementation (Follitropin alpha) in patients aged ≥ 35 years undergoing IVF treatment.

Study hypothesis: Pergoveris (LH supplementation) is better than follitropin alpha (non-LH supplementation) for ovarian stimulation in aged IVF patients.

DETAILED DESCRIPTION:
A randomized controlled single center study.

Based on the difference of 19.1% in the clinical pregnancy rate between the two treatment groups, with and without LH supplementation, in a previous study, with 90% power and a 2-sided P-value of 0.05, the number of subjects required was 109 per group (total 218). The recruitment target was 120 subjects per group (total 240) to allow for dropouts.

Eligible subjects were randomized in blocks of 4 via a computer generated random number list to either the Pergoveris arm or the follitropin alpha arm.

Ovarian stimulation was performed by using GnRH antagonist protocol.

Follitropin alfa (recombinant FSH) was administered on day 2 or day 3 of the menstrual cycle. The first FSH dose was determined according to each individual patient, based on the process as follows:

* AFC ≤ 6: 300 IU/day
* AFC 7-15: 225 IU/day
* AFC ≥ 16: 150 IU/day

GnRH antagonist (Cetrotide, Merck-Serono) was administered on day 5 of FSH administration.

* Recombinant LH (in the form of Pergoveris) was supplemented from day 6 of FSH administration. Patients in the Pergoveris group would be administered a reduced dose of recombinant FSH (reduced by 150 IU/day) which was replaced with Pergoveris (150IU FSH + 75IU LH)/day.
* The Follitropin alpha group retained recombinant FSH. In both groups, if the number of developing follicles was inappropriate, the dose could be titrated depending on the physician's judgment.

Monitoring the follicular development was performed by vaginal ultrasound probe, quantifying LH, estradiol and progesterone, starting from day 5 of FSH, based on the current processes of the hospital.

OPU and embryo transfer: OPU was performed 36 hours after hCG administration. Embryos were transferred on day 2.

Luteal phase support: daily vaginal progesterone

Pregnancy testing and ultrasound: a pregnancy test was done 14 days after embryo transfer. Beta hCG > 5mIU/ml was considered positive. Fetal ultrasound was performed 3 weeks after a positive pregnancy test to verify clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 35 years
* body mass index <28 kg/m2
* had ≤ 3 previous IVF attempts
* receiving a GnRH-antagonist protocol
* agreement to participate in the study, and to disclose any medical events to the investigator. The subject must be willing and able to comply with the protocol requirements for the duration of the study.
* have given written informed consent with the understanding that the subject may withdraw consent at any time

Exclusion Criteria:

* participating in another interventional clinical trial
* PCOS or WHO group 1
* have uterine abnormalities
* have endocrine disorders such as hyperprolactinemia, thyroid disorders

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 7 weeks after embryo transfer
  Clinical pregnancy is defined by the image gestational sac under ultrasonography.
Live birth | at the time of delivery
  Live birth is defined if a live newborn delivered.

SECONDARY OUTCOMES:
Total FSH international units (IU) used for stimulation | Measure at the time when stimulation finishes, eg. in average 10-11 days, maximum 20 days
  Calculate total number of IU of FSH used for stimulation at the last day of stimulation regime.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — CGRH, School of Medicine, Vietnam National University HCMC, Vietnam
Locations (1):
- An Sinh Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Vuong TN, Phung HT, Ho MT. Recombinant follicle-stimulating hormone and recombinant luteinizing hormone versus recombinant follicle-stimulating hormone alone during GnRH antagonist ovarian stimulation in patients aged >/=35 years: a randomized controlled trial. Hum Reprod. 2015 May;30(5):1188-95. doi: 10.1093/humrep/dev038. Epub 2015 Mar 3. PMID 25740882